CLINICAL TRIAL: NCT05146102
Title: Ethics Communication in Groups Among Healthcare Professionals (The Ethics-com Study).
Acronym: Ethics-com
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Margareta Brännström, professor, Umeå University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ethics-com001
Record Dates: First submitted 2021-11-05; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Ethics Support
Keywords: ethics support; ethical rounds; healthcare personnel
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The interventiongroup is offered organized interprofessional sessions, once a month, for six months at their workplace. In the the controlgroup, organized interprofessional sessions are not planned at the wards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ethics communication in group, in line with "the one to five-step method" (Experimental): Healthcare professionals working as "ethical representatives" at the current ward (n=5) have recently gone through a basic ethics program. They will continue by going through an education program for facilitating ethics communication in group, in line with "the one to five-step method"
  * The education program has a theoretical and practical approach, which includes the theoretical base of the ethical communication in groups and practicing "the one to five method"
  * Thereafter, each "ethical representative" will facilitate interprofessional sessions at a clinical ward, once a month, for six months at their workplace. Gathering meetings for feedback will be offered for the "ethical representatives" once a month.
  Interventions: Other: ethics communication in group, in line with "the one to five-step method"
- No organized ethics communication in group (No Intervention): Healthcare professionals working as "ethical representatives" at the current ward (n=5) have recently gone through a basic ethics program. They have not being educated in "the one to five-step method and organized interprofessional sessions are not planned at the wards.

INTERVENTIONS:
Other: ethics communication in group, in line with "the one to five-step method" — Healthcare professionals working as "ethical representatives" at the current ward (n=5) have recently gone through a basic ethics program. They will continue by going through an education program for facilitating ethics communication in group, in line with "the one to five-step method"
  The education program has a theoretical and practical approach, which includes the theoretical base of the ethical communication in groups and practicing "the one to five method" Thereafter, each "ethical representative" will facilitate interprofessional sessions at a clinical ward, once a month, for six months at their workplace. Gathering meetings for feedback will be offered for the "ethical representatives" once a month.
  Arms: ethics communication in group, in line with "the one to five-step method"

SUMMARY:
Moral distress has been described as a condition with frustration, guilt, anger and as one reason for health care professionals to leave the profession. Ethics communication in groups has been showed to work as support for health care professionals in ethically difficult situations and further work as a tool to improve the ethical climate and prevent moral distress. Our research group has developed the "one to five-step method" for interprofessional ethical communication in groups. The overall aim of this project: is to implement and evaluate a method for organized interprofessional communication about ethical issues in healthcare.

DETAILED DESCRIPTION:
Ethically difficult situations are a part of the everyday clinical practice for health care professionals and concerns difficult judgements, prioritization and crucial decisions. Being unable or prevented to act according to one's moral conviction for what is good and right care may increase the risk for health care professionals to experience moral distress. Moral distress has been described as a condition with frustration, guilt, anger and as one reason for health care professionals to leave the profession. Ethics communication in groups has been showed to work as support for health care professionals in ethically difficult situations and further work as a tool to improve the ethical climate and prevent moral distress. Our research group has developed the "one to five-step method" for interprofessional ethical communication in groups. The method is a stepwise support for facilitating ethics communication in clinical practice when the situations occurs. The overall aim of this project: is to implement and evaluate a method for organized interprofessional communication about ethical issues in healthcare.

Significance: The study can generate knowledge about ethics communication in groups in line with the " one to five step method", reduce moral distress, create improved ethical climate for healthcare professionals and in turn open up prerequisites for good care.

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals working at included wards

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
moral distress meausered by using the Meausure of Moral Distress for Health care Professionals (MMD-HP) and the Moral Distress Thermometer | Change from Baseline moral distress at 6 months
  primary outcome

SECONDARY OUTCOMES:
ethical climate meausered by the Swedish ethical climate questionnaire (SwECQ) | Change from Baseline ethical climate at 6 months
  secondary outcome
experiences | at 6 month
  interviews of the interventiongroup

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Brännström, Principal Investigator — Umea university, department of nursing, Umeå, Sweden
Locations (2):
- Sweden (2):
  - Margareta Brännström, Skellefteå, Umeå Universitet
  - Umeå university, Umeå, Umeå Universitet

REFERENCES:
- [Derived] Margareta B, Ulf I, C FG. Effects of ethics communication in health care: a cluster randomised controlled trial. BMC Med Ethics. 2025 Jul 26;26(1):106. doi: 10.1186/s12910-025-01270-w. PMID 40713613